CLINICAL TRIAL: NCT04854915
Title: Mobile Health Biometrics to Enhance Exercise and Physical Activity Adherence in Children and Young People With Obesity
Brief Title: mHealth Biometrics for Young People With Obesity (MOTIVATE- LOOP)
Acronym: MOTIVATE-L
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liverpool John Moores University (Other)
Collaborators: Alder Hey Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MOTIVATE- LOOP
Record Dates: First submitted 2021-04-06; First posted 2021-04-22 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-04

CONDITIONS: Obesity, Adolescent
Keywords: mobile health technology; physical activity; exercise; exercise prescription/ education; exercise adherence
MeSH Terms: conditions — Pediatric Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: pilot, parallel group, randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liverpool Overweight and Obesity Programme (LOOP) only (Active Comparator): Patients will continue to follow the LOOP@ Alder Hey programme.
  Interventions: Behavioral: LOOP Only
- LOOP + mHealth technology assisted exercise counselling (Experimental): Patients will continue to work with the LOOP MDT. However, exercise and physical activity advise will be taken over by an exercise specialist. Participants will co-develop a 3-month structured exercise and PA programme, with support from an exercise specialist. All participants will have 5 exercise consultations with their exercise specialist. The intervention will be supported by 3 mHealth elements; 1) a wrist worn fitness watch, 2) a smartphone app for patients, and 3) a coaching website for the exercise specialist. The 3 elements will be synced, allowing data to be transferred between platforms.
  Interventions: Behavioral: LOOP + mHealth technology assisted exercise counselling

INTERVENTIONS:
Behavioral: LOOP + mHealth technology assisted exercise counselling — Participants will complete a 3 month exercise and physical activity intervention supported by mHealth technology
  Arms: LOOP + mHealth technology assisted exercise counselling
Behavioral: LOOP Only — Participants will complete the LOOP @ Alder Hey programme
  Arms: Liverpool Overweight and Obesity Programme (LOOP) only

SUMMARY:
The investigators aim to undertake a feasibility randomised controlled trial (RCT) to investigate whether mHealth technology, allowing biometric informed feedback and coaching on exercise and PA, can be incorporated into the existing Liverpool Overweight and Obesity Programme (LOOP) at Alder Hey Children's Hospital. The overall objective is to have an evidence-based exercise and PA intervention ready to evaluate in a future RCT.

DETAILED DESCRIPTION:
The study will recruit patients from the Liverpool Overweight and Obesity Programme at Alder Hey Children's Hospital (LOOP@ Alder Hey). 40 participants will be recruited and randomly assigned to one of two groups (Control n=20, Intervention n=20). Patients in the control group will continue to follow the LOOP@ Alder Hey programme but physical activity sessions will be monitored during the 12-week intervention using a heart rate monitor. Importantly, the heart rate monitor will not provide any feedback to the patient. The intervention group will be provided with exercise counselling and to support this they will also be provide with a wristwatch that can monitor everyday activity and their heart rate, a smartphone app and access to a website. The intervention group will also participate in 5 consultations with an exercise specialist to plan their exercise programme and be updated on their progress towards physical activity targets. Weekly text message updates will also provide feedback to the intervention group with participants able to respond to these updates. Before and after the 3-month supported interventions, volunteers will participate in testing to assess changes in physical activity, blood pressure, glycaemia control, body composition and health related quality of life. Interviews with participants, parents and the LOOP Clinic multidisciplinary team will form the basis for a review of the pilot randomised control trial. Participants will also fill out 6 validated questionnaires about motivations, the impact of their condition on daily life and their typical exercise levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients within the Liverpool Overweight and Obesity Programme aged 12-18 years
* BMI>30
* Receiving input from members of LOOP clinic at Alder Hey for weight management
* For those prescribed Metformin: Stable dose for 3-months or more

Exclusion Criteria:

* Severe learning/behaviour difficulties
* Severe autism
* Secondary causes of obesity like Cushing's disease
* Syndromic causes of obesity
* Patients on GLP-1 analogues for obesity
* Type 2 diabetes mellitus
* Require an interpreter

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Through study completion, an average 16 weeks
  Determine the number of young people referred to the LOOP that are eligible to participate, the proportion of these who would be willing to take part in this trial (i.e., recruitment rate), and their characteristics
Drop out | Through study completion, an average 16 weeks
  Determine the number of young people retained at 3-months (i.e., participant drop-out).

SECONDARY OUTCOMES:
Device derived adherence to structured exercise | Up to 12 weeks
  Number of exercise sessions per week
Device derived duration of exercise | Up to 12 weeks
  minutes of exercise completed per session
Device derived intensity of structured exercise | Up to 12 weeks
  intensity of exercise sessions performed (percentage of HR max)
Device derived physical activity (GENEActiv) | Baseline and the final 2 weeks of the intervention (weeks 10-12)
  Minutes of low, moderate and vigorous physical activity
Survey reported exercise behaviour | Baseline, 4 and 8 weeks into the intervention and immediately after the intervention
  Bouts of mild, moderate and strenuous exercise lasting ≥30 minutes
Height | Baseline and immediately after the intervention
  Height (m)
Weight (kg) | Baseline and immediately after the intervention
  Weight (kg)
Body composition | Baseline and immediately after the intervention
  bioimpedence (fat mass (and lean mass)
Blood pressure | Baseline and immediately after the intervention
  Blood pressure (systolic and diastolic)
Concentration of Hba1c | Baseline and immediately after the intervention
  Hba1c
Fasted insulin concentration | Baseline and immediately after the intervention
  Fasted insulin
Fasted glucose concentration | Baseline and immediately after the intervention
  Fasted glucose
Glycaemic control | Baseline and the final 2 weeks of the intervention (weeks 10-12)
  Flash glucose monitoring
Blood Lipid concentrations | Baseline and immediately after the intervention
  Total cholesterol, HDL/LDL, Triglycerides
Liver function concentrations | Baseline and immediately after the intervention
  AST, ALT, Albumin
C-peptide concentration | Baseline and immediately after the intervention
  C-peptide
Health related quality of life as assessed by the PedsQL 4.0 | Baseline and immediately after the intervention
  Paediatric Quality of Life Inventory (PedsQL) 4.0 Max score 115, min score 0, high score is better
Health related quality of life as assessed by the EQ-5D-Y | Baseline and immediately after the intervention
  EuroQol- 5 Dimension Youth version (EQ-5D-Y), Max score 15, min score 5, high score is better
Health related quality of life as assessed by the KIDSCREEN-52 | Baseline and immediately after the intervention
  KIDSCREEN-52. Max score 260, min score 52, high score is better
Exercise motivation | Baseline and immediately after the intervention
  Behavioural regulation in exercise questionnaire-2 (BREQ-2). Max score 76, min score 0, high score is better
Patient Interview to access intervention acceptability | Within 2 weeks of the end of the intervention
  Patient interview
Parent Interview to access intervention acceptability | Within 2 weeks of the end of the intervention
  Parent interview
multidisciplinary team focus group to assess intervention acceptability | 1 year
  Focus group with multidisciplinary LOOP team
Process evaluation | Within 2 weeks of the end of the intervention
  Participant interview

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Liverpool John Moores University, Liverpool
  - Alder Hey Childrens NHS Foundation Trust, Liverpool

IPD SHARING:
Plan to Share IPD: No
No plan to share